CLINICAL TRIAL: NCT04899713
Title: Long-term Survival of Locally Advanced Breast Cancer Patients Treated With Neoadjuvant Chemotherapy With or Without Zoledronic Acid (ZOMETA®)
Brief Title: NEOZOL_Follow-up Study
Acronym: NEOZOL_FU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0552
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Locally Advanced Breast Cancer
Keywords: Breast cancer; Zometa®; Survival survey; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group (neo-adjuvant chemotherapy combined with ZOMETA®) (zoledronic acid): Patients treated every 3 weeks (+/- 2 days ) for 8 cycles in total. The 4 first cycles : zoledronic acid 4 mg (in a 15 min. infusion) + doxorubicin (60 mg/m²) + cyclophosphamide (600 mg/m²). The 4 last cycles with zoledronic acid 4 mg (in a 15 min. infusion) + docetaxel (100 mg/m²)
  Interventions: Other: Survival survey
- Control group (neo-adjuvant chemotherapy alone): Patients treated every 3 weeks (+/- 2 days) for 8 cycles in total. The 4 first cycles : doxorubicin (60 mg/m²) combined with cyclophosphamide (600 mg/m²). The 4 last cycles with docetaxel (100 mg/m²)
  Interventions: Other: Survival survey

INTERVENTIONS:
Other: Survival survey — To assess the effect of adding ZOMETA® to neoadjuvant chemotherapy on event-free survival.

SUMMARY:
Breast cancer is the most common cancer in women and is the leading cause of death from cancer in France.

The main types of treatment used to treat breast cancer are surgery, chemotherapy, radiotherapy, hormone therapy and targeted therapies. In locally advanced breast cancer, a neo-adjuvant chemotherapy treatment is currently recommended as it may provide a sufficient tumour response to allow for conservative breast treatment.

Zoledronic acid (ZOL) is an N-biphosphonate used in the prevention of bone complications and in the treatment of hypercalcaemia In vitro and in vivo studies have shown an effect of ZOL on tumour and endothelial cells, supporting an anti-tumour activity of N-biphosphonates.

Between April 2010 and October 2013, 50 patients with locally advanced breast cancer were randomized in the NEOZOL study to receive neoadjuvant chemotherapy with (n=26) or without (n=24) zoledronic acid (ClinicalTrials.gov Identifier: NCT01367288). The primary objective of this study was to evaluate the effect of the addition of ZOMETA® to neoadjuvant chemotherapy on the change in serum VEGF concentration before and after neoadjuvant treatment (i.e. at the time of surgery).

Assessment of long-term survival was not planned in the NEOZOL study protocol. The objective of NEOZOL_FU study is to evaluate the survival of patients included in the NEOZOL study, 7 years after inclusion of the last patient.

This study will provide essential data on the long-term survival and risk of relapse of patients with locally advanced breast cancer who have received neo-adjuvant chemotherapy with or without zoledronic acid (ZOMETA®).

ELIGIBILITY:
Inclusion Criteria:

* Woman who signed a written consent, included and randomised in the main analysis of the NEOZOL study

Exclusion Criteria:

* Patient's opposition to the use of her data in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 50 patients with locally advanced breast cancer (TNM IIa or IIb or IIIa, tumor > 2 cm, ductal or lobular histology), who benefited from neoadjuvant chemotherapy associated ( n = 26) or not (n = 24) with the zoledronic acid, and having participated in the NEOZOL study (NCT01367288)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 31/12/2019
  Event-free survival is defined as the time between the date of randomization and the date of the 1st event among: 1st documented locoregional or metastatic infiltrating relapse (not including in situ relapses) or death from whatever cause.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Centre hospitalier de Bourg en Bresse, Hôpital Fleyriat, Service d'Onco-Hématologie et de Gynécologie Obstétrique, Bourg-en-Bresse
  - Hôpital Femme Mère Enfant, Groupement Hospitalier EST, Service de Gynécologie Clinique, Bron
  - Centre de Lutte Contre le Cancer - Institut Jean Perrin, Service de Médecine Oncologique, Clermont-Ferrand
  - Centre Hospitalier Alpes Léman, Service de Gynécologie, Contamine-sur-Arve
  - Centre Hospitalier Universitaire de Limoges, Hôpital Dupuytren 1, Service d'Oncologie Médicale,, Limoges
  - Centre Léon Bérard, Département de Cancérologie Médicale, Lyon
  - Hôpital Européen, Service d'Oncologie, Marseille
  - Centre Hospitalier Universitaire de Montpellier - Hôpital St Eloi, Montpellier
  - Centre Hospitalier Universitaire de Poitiers, Hôpital la Milétrie, Poitiers
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Hospitalier de Thonon Hôpitaux du Léman, site Georges Pianta Service de Gynécologie Obstétrique, Thonon-les-Bains